CLINICAL TRIAL: NCT00532480
Title: Duloxetine Effects on Brain fMRI Response to Emotionally Valenced Pictures in the Treatment of Patients With Major Depression
Brief Title: Study of Brain Response to Emotional Pictures Using a fMRI While on Duloxetine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0607-22
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Major Depression
Keywords: Depression; Duloxetine; fMRI; pictures
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duolxetine (Other): Open-label duloxetine 30 - 60 mg oral administration
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — 60 mg capsules
  Other Names: Cymbalta

SUMMARY:
The purpose of this study is to find out what parts of the brain have increased or decreased activity when people are depressed and how antidepressant medicine changes this activity in depressed patients. The genetic samples collected are to look at variation in a gene (serotonin transporter gene), which affects the functioning of the chemical serotonin in the brain

DETAILED DESCRIPTION:
This study will measure the activity in different parts of the brain, while the patients are seeing some pictures, using Magnetic Resonance Imaging (MRI) scan. For this study three MRI scans will be conducted. One before the patient begins on any medication, one during the study after 3 weeks of treatment and one after six more weeks of treatment with a standard antidepressant called duloxetine.

ELIGIBILITY:
Inclusion Criteria for Depressed Patients:

* Ages 18 - 60 years and able to give voluntary informed consent.
* Satisfy criteria for Major Depressive Disorder (MDD) and current depressed episode using the Structured Clinical Interview for DSM-IV (SCID-IV).
* 17-item Hamilton Depression Rating Scale (HDRS) score > 18.
* Satisfy criteria to undergo an MRI scan based on MRI screening questionnaire.
* Able to be managed as outpatients for initial assessment and during treatment as ascertained by the following:

  * Symptoms not worsening by more than 10 points on the HDRS during the course of the study.
  * No danger to self or others.

Exclusion criteria for patients:

* Meeting DSM-IV criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, bipolar disorder, atypical psychosis, mental retardation, or organic mental (including organic mood) disorder.
* Known hypersensitivity to duloxetine or any of the inactive ingredients.
* On monoamine oxidase inhibitors in the past 2 weeks.
* History of narrow angle glaucoma
* Lack of response of the current episode of depression to two or more adequate courses of antidepressant therapy at a clinically appropriate dose for a minimum of 4 weeks or, in the judgment of the investigator, the patient meets criteria for treatment-resistant depression.
* Use of neuroleptic in the past 2 weeks.
* Use of antidepressants in the past 2 weeks. If on fluoxetine in the past, then should not have been on this medication for 4 weeks.
* History of lack of response to duloxetine.
* Use of mood stabilizers in the past 2 weeks.
* Use of benzodiazepines in the past 2 weeks.
* Acutely suicidal or homicidal or requiring inpatient treatment.
* Meeting DSM-IV criteria for other substance dependence within the past year, except caffeine or nicotine. The criteria will be evaluated by interview and urinary toxicology screening initially and on test days.
* Use of alcohol in the past 1 week.
* No serious medical or neurological illness as assessed by physical examination and laboratory examination including CBC and blood chemistry.
* Current pregnancy or breast-feeding.
* Metallic implants.
* Previously known positive HIV blood test as reported by the subject.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — Indiana University Schoole of Medicine
Locations (1):
- Indiana University Adult Psychiatric Clinic, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Duloxetine: Duloxetine 60 mg capsules orally daily open label
Period: Overall Study
Arm/Group | Duloxetine
Started | 10
Completed | 7
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine: Duloxetine : 60 mg capsules
Arm/Group | Duloxetine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: 17-item Hamilton Depression Rating Scale
Description: Standard 17-item rating scale for depression used in clinical trials. A score of 0-7 is considered to be normal. 8 - 13 mild depression. Scores of 20 or higher indicate moderate, severe, or very severe depression, and are usually required for entry into a clinical trial. Range of score: 0 - 50.
Time Frame: 8 weeks
Population: 10 patients included in the study out of which 7 completed 8 weeks of the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 7
units on a scale
  Baseline 17-item HDRS | 19 (5)
  Post-treatment 17-item HDRS | 10 (5)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=10)
decreased libido (Nervous system disorders) | 4 (4)
headache (Nervous system disorders) | 3 (3)
Irritability (Psychiatric disorders) | 3 (3)
tremor (Nervous system disorders) | 2 (2)
increased appetite (Metabolism and nutrition disorders) | 2 (2)
crying more often (Psychiatric disorders) | 1 (1)
indigestion (Gastrointestinal disorders) | 1 (1)
panic attack (Psychiatric disorders) | 1 (2)
sweating (Nervous system disorders) | 1 (1)
flushing (Nervous system disorders) | 1 (1)
nervousness (Psychiatric disorders) | 1 (1)
no orgasm (Nervous system disorders) | 1 (1)
premature ejaculation (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No